CLINICAL TRIAL: NCT01371669
Title: Study Searching for Hypoxemic Sleep Breathing Disorders in a Cohort of Patients With Idiopathic Pulmonary Arterial Hypertension (IPAH) and Chronic Post-embolic Pulmonary Hypertension (CPEPH)
Brief Title: Screening for Sleep Hypoxemia in Pulmonary Arterial Hypertension
Acronym: Sommeil_HTAP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P090206
Record Dates: First submitted 2010-12-13; First posted 2011-06-13 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Sleep Disorders
Keywords: Pulmonary arterial hypertension; Chronic post embolic disease; Sleep hypoxemia; polysomnography; sleep apnea; periodic respiration
MeSH Terms: conditions — Sleep Wake Disorders; Pulmonary Arterial Hypertension; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IPAH or CPEPH: Idiopathic pulmonary arterial hypertension (IPAH) or pulmonary hypertension associated with chronic post-embolic pulmonary hypertension (CPEPH)

SUMMARY:
In the investigators study, and regarding results of small cohorts in the literature, the investigators hypothesize that hypoxemia is frequent in IPAH and CPEPH. The investigators will explore these patients with a one night polysomnography and transcutaneous capnography, searching for hypoxemia and hypercapnia and by determining its physiopathologic mechanisms.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is a rare and severe disease of young adults, characterized by a progressive increase in pulmonary vascular resistances leading to cardiac failure and death. Patients with PH are categorized in two major groups: primary PH (PPH) wich is idiopathic, and secondary PH associated with many conditions such as chronic pulmonary embolic diseases (CPED).Increase in vascular resistance in PH is secondary to vasoconstriction and to a proliferative remodeling process of the arterial wall leading to obliteration of the small arterioles. On the other hand, hypoxemia is known to cause similar changes in vascular architecture. Also, some small cohorts study in the literature mentioned an increase of sleep hypoxemia prevalence accounting for almost 70% of cases. The mechanisms of this hypoxemia are completely unknown.Our study is observational, prospective and transversal, searching for hypoxemic respiratory sleep disorders (HRSD) in PPH and in CPEPH. Included patients will have one night polysomnography (CIDELEC) with a continuous measurement of transcutaneous PCO2.The major objectives are to determine the prevalence of HRSD, their physiopathologic mechanisms and their possible causal factors according to PH history, clinical findings and hemodynamic severity.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 75 years
* Patient with IPAH ot CPEPH stable for at least 3 months. Stability is defined by the New York Heart Association classes for dyspnea and the six minutes walking test (6MWT). Furthermore, no changes in medical therapy had occured during the last three months.
* Patients who signed informed consent

Exclusion Criteria:

* Patients with secondary PH associated with other pathologies outside CPEPH ( sclerodermia, systemic lupus erythematous, portal hypertension, chronic HIV infection...)
* Patients who had a functional and/or a hemodynamic degradation during the last 3 months or a change in pulmonary hypertension treatment
* Patients with obstructive or restrictive ventilatory disorder with a Ventricular Ejection Fraction <60% predicted
* Women without effective contraception
* Patients with a Body Mass Index above 35 kg/m2
* Patient not affiliated to a social security scheme

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with IPAH or CPEPH hospitalized in our pulmonary department for a standard follow-up. They have to be in a stable condition, as defined by the New York Heart Association classes for dyspnea and the six minutes walking test. Furthermore, no changes in medical therapy could have been made during the last three months.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
hypoxemia during the night | at the inclusion
  prevalence of nocturnal hypoxemia in IPAH and CPEPH

SECONDARY OUTCOMES:
Predictors: physical, functional and hemodynamical data | at the inclusion
  Predictive factors of sleep hypoxemia in IPAH and CPEPH
Physiopathologic mechanisms: causes of nocturnal hypoxemia: hypoventilation, sleep disordered breathing, shunting, V/Q mismatch | at the inclusion
  Physiopathologic mechanisms of sleep hypoxemia in IPAH and CPEPH

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel ROISMAN, MD, Principal Investigator — Assistance Publique - Hopitaux de Paris, Hôpital Antoine Beclere
Locations (1):
- Assistance Publique- Hôpitaux de Paris: Antoine Beclere Hospital, Clamart, France

REFERENCES:
- [Derived] Jilwan FN, Escourrou P, Garcia G, Jais X, Humbert M, Roisman G. High occurrence of hypoxemic sleep respiratory disorders in precapillary pulmonary hypertension and mechanisms. Chest. 2013 Jan;143(1):47-55. doi: 10.1378/chest.11-3124. PMID 22878784